CLINICAL TRIAL: NCT00514709
Title: Immunogenicity Study of the Antibody Persistence and Booster Effect of DTaP-Hep B-PRP-T Combined Vaccine at 12 to 18 Months of Age Following a Primary Series at 6, 10 and 14 Weeks of Age in Healthy Filipino Infants Having Received Hepatitis B Vaccine at Birth
Brief Title: Immunogenicity Study of Antibody Persistence and Booster Effect of DTaP-HB PRP~T Combined Vaccine in Filipino Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AL204
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Results first posted 2013-11-14 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Influenza
Keywords: Diphtheria; Tetanus; Pertussis; Hepatitis B Hansenula (HB); Haemophilus influenzae type b
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Influenza, Human; Haemophilus Infections | interventions — diphtheria-tetanus-acellular pertussis-Hib-hepatitis B vaccine; Poliovirus Vaccine, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): DTaP-Hep B-PRP-T + OPV vaccine group
  Interventions: Biological: DTaP-HB PRP~T Combined Vaccine; Biological: Oral Polio Vaccine
- Group 2 (Experimental): Tritanrix-HepB/Hib™ + OPV vaccine group
  Interventions: Biological: DTaP-HB-PRP~T vaccine; Biological: Oral Polio Vaccine

INTERVENTIONS:
Biological: DTaP-HB PRP~T Combined Vaccine — 0.5 mL, Intramuscular (IM)
  Arms: Group 1
Biological: DTaP-HB-PRP~T vaccine — 0.5 mL, IM
  Arms: Group 2
Biological: Oral Polio Vaccine — Oral co-administered with study vaccine.

SUMMARY:
DTaP-HB-PRP~T combined vaccine is being developed in order to comply with expanding programs for immunization in infancy, while offering the benefit of a reduced number of injections, and potentially of an increased acceptance.

Primary Objectives:

* To describe the antibody persistence at 12 to 18 months following a three-dose primary series vaccination of either DTaP-HB-PRP~T or Tritanrix-Hep B/Hib™ given at 6, 10 and 14 weeks of age, and one dose of Hepatitis B (Hep B) vaccine given at birth.
* To describe the effect of a booster dose of DTaP-HB-PRP~T on immunogenicity at 12 to 18 months following a three-dose primary series vaccination of either DTaP-HB-PRP~T or Tritanrix HepB/Hib™ given at 6, 10 and 14 weeks of age, and one dose of Hep B vaccine given at birth.

Secondary Objective:

* To describe the safety profile of the booster dose of the DTaP-HB-PRP~T vaccine when administered concomitantly with Oral Polio Vaccine (OPV).

DETAILED DESCRIPTION:
This study will assess the immunogenicity and reactogenicity of the investigational DTaP-HB-PRP~T combined vaccine when given as a booster dose, concomitantly with OPV, in Filipino children previously primed at 6, 10, and 14 weeks with the investigational DTaP-HB-PRP~T combined vaccine or Tritanrix-Hep B/Hib™ vaccine and having received a first dose of Hep B vaccine (Recomvax B™) at birth in a previous study, AL201 (NCT00348881).

ELIGIBILITY:
Inclusion Criteria:

* Toddler aged 12 to 18 months of age on the day of inclusion (range: 365 days to 578 days of age inclusive)
* Participated in the AL201 study and completed the three-dose primary series with either DTaP-HB-PRP~T or Tritanrix-HepB/Hib™, and OPV, at 6, 10 and 14 weeks of age, and received hepatitis B vaccine at birth
* Informed consent form signed by one parent or legal representative if appropriate (independent witness mandatory if parent is illiterate)
* Able to attend all scheduled visits and to comply with all trial procedures

Exclusion Criteria:

* Participation in another clinical trial in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term (for more than 2 weeks) systemic corticosteroid therapy within the preceding 3 months
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to a vaccine containing the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion
* Blood or blood-derived products received in the last 3 months
* Any vaccination in the 4 weeks preceding the trial vaccination
* Vaccination planned in the 4 weeks following the trial vaccination
* Febrile (temperature ≥ 38.0°C) or acute illness on the day of inclusion
* History of documented diphtheria, tetanus, pertussis, Haemophilus influenzae type b, hepatitis B or poliomyelitis infection(s) (confirmed either clinically, serologically, or microbiologically)
* Vaccination with a vaccine containing diphtheria, tetanus, pertussis, Haemophilus influenzae type b, hepatitis B or poliovirus 3 types antigen, since the end of the primary series
* Thrombocytopenia or a bleeding disorder contraindicating IM vaccination
* Serious adverse event related to any vaccination in the AL201 study.

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1843 (Actual)
Dates: Start 2007-09; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (7):
- Philippines (7):
  - City of Muntinlupa, Alabang Junction Alabang
  - City of Muntinlupa, Alabang
  - City of Muntinlupa, Bayanan Annex
  - City of Muntinlupa, Cupang
  - City of Muntinlupa, Filinvest
  - City of Muntinlupa, Putatan
  - City of Muntinlupa, Tunasan

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized and enrolled from 06 August 2007 to 29 July 2008 in 2 clinic centers in the Philippines.
Pre-assignment Details: A total of 1843 participants who met all the inclusion and none of the exclusion criteria were enrolled and vaccinated.
Groups:
- Group 1: DTaP-Hep B-PRP~T + OPV: Participants received a booster dose of the DTaP-Hep B-PRP~T Combined vaccine concomitantly with oral polio vaccine (OPV) following a 3-dose primary series of DTaP-Hep B-PRP~T combined vaccine concomitantly with OPV at 6, 10, and 14 weeks of age in Study AL201 (NCT00348881).
- Group 2: Tritanrix-Hep B/ Hib™ + OPV: Participants received a booster dose of the DTaP-Hep B-PRP~T Combined vaccine concomitantly with oral polio vaccine (OPV) following a 3-dose primary series of Tritanrix-Hep B/Hib™ concomitantly with OPV at 6, 10, and 14 weeks of age in Study AL201 (NCT00348881).
Period: Overall Study
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Started | 1230 | 613
Completed | 1230 | 613
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: DTaP-Hep B-PRP~T + OPV: Participants received a booster dose of the DTaP-Hep B-PRP~T Combined vaccine concomitantly with oral polio vaccine (OPV) following a 3-dose primary series of DTaP-Hep B-PRP~T combined vaccine concomitantly with OPV at 6, 10, and 14 weeks of age in Study AL201.
- Group 2: Tritanrix-Hep B/ Hib™ + OPV: Participants received a booster dose of the DTaP-Hep B-PRP~T Combined vaccine concomitantly with oral polio vaccine (OPV) following a 3-dose primary series of Tritanrix-Hep B/Hib™ concomitantly with OPV at 6, 10, and 14 weeks of age in Study AL201.
- Total: Total of all reporting groups
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV | Total
Number analyzed (Participants) | 1230 | 613 | 1843
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1230 | 613 | 1843
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 15.1 (1.96) | 15.1 (1.95) | 15.1 (1.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 629 | 302 | 931
  Male | 601 | 311 | 912
Region of Enrollment [Number; unit: Participants]
  Philippines | 1230 | 613 | 1843

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Antibody Persistence and Immunogenicity Booster Response to Vaccination With DTaP-Hep B-PRP~T Concomitantly With Oral Polio Vaccine (OPV)
Description: Immunogenicity was assessed by means of radioimmunoassay (RIA) for anti-Hepatitis B (Hep Bs) and anti-PRP antibodies, enzyme immunoassay (EIA) for anti-Tetanus, and serum neutralization (SN) for anti-Diphtheria.
  Booster responses defined as titers ≥ 10 mIU/mL for anti-Hep Bs; ≥ 0.15 μg/mL for anti-PRP; ≥ 0.01 IU/mL for anti-Tetanus and anti-Diphtheria; Pertussis Toxoid and Filamentous Hemagglutinin (FHA) 4-fold increase and booster response.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-booster vaccination
Population: Antibody persistence and immunogenicity booster responses were assessed in a subset of participants available for the endpoint, the per-protocol population.
Measure: Number; unit: Participants
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Number analyzed (Participants) | 93 | 105
Participants
  Anti-Hep B Pre-booster (N = 93, 103) | 81 | 80 [0 to 0]
  Anti-Hep B Post-booster (N = 93, 105) | 91 | 103
  Anti-PRP Pre-booster (N = 93, 105) | 78 | 105 [0 to 0]
  Anti-PRP Post-booster (N = 93, 105) | 93 | 105
  Anti-Diphtheria Pre-booster (N = 93, 105) | 72 | 68 [0 to 0]
  Anti-Diphtheria Post-booster (N = 93, 105) | 93 | 103
  Anti-Tetanus Pre-booster (N = 93, 105) | 93 | 105 [0 to 0]
  Anti-Tetanus Post-booster (N = 93, 105) | 93 | 105
  Anti-Pertussis 4-Fold increase (N = 89, 101) | 85 | 100
  Anti-Pertussis booster response (N = 89, 101) | 87 | 101
  Anti-FHA 4-Fold increase (N = 91, 103) | 80 | 102
  Anti-FHA booster response (N = 91, 103) | 89 | 102

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Vaccine Antibodies After Booster Vaccination With DTaP-Hep B-PRP~T Combined Vaccine Concomitantly With Oral Polio Vaccine (OPV)
Description: Immunogenicity was assessed by means of radioimmunoassay (RIA) for anti-Hepatitis B (Hep Bs) and anti-PRP antibodies, enzyme immunoassay (EIA) for anti-Tetanus, and serum neutralization (SN) for anti-Diphtheria following the booster vaccination.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: GMTs were assessed in a sub-set of the participants available for the endpoint, the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Group 1: DTaP-Hep B-PRP-T + OPV: Participants received a booster dose of the DTaP-Hep B-PRP~T Combined vaccine following a 3-dose primary series of DTaP-Hep B-PRP-T combined vaccine concomitantly with OPV at 6, 10, and 14 weeks of age in Study AL201.
- Group 2: Tritanrix-Hep B/ Hib™ + OPV: Participants received a booster dose of the DTaP-Hep B-PRP~T Combined vaccine following a 3-dose primary series of Tritanrix-Hep B/ Hib™ concomitantly with OPV at 6, 10, and 14 weeks of age in Study AL201.
Arm/Group | Group 1: DTaP-Hep B-PRP-T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Number analyzed (Participants) | 93 | 105
Titers
  Anti-Hep B Pre-booster (N = 93, 103) | 71.6 [51.1 to 100] | 42.2 [30.5 to 58.5]
  Anti-Hep Bs Post-booster (N = 93, 105) | 4224 [2760 to 6464] | 3673 [2441 to 5527]
  Anti-PRP Pre-booster (N = 93, 105) | 0.889 [0.602 to 1.31] | 5.32 [4.13 to 6.84]
  Anti-PRP Post-booster (N = 93, 105) | 58.1 [40.4 to 83.4] | 242 [195 to 299]
  Anti-Diphtheria Pre-booster (N = 93, 105) | 0.016 [0.013 to 0.021] | 0.014 [0.011 to 0.018]
  Anti-Diphtheria Post-booster (N = 93, 105) | 1.36 [1.05 to 1.77] | 1.43 [1.06 to 1.93]
  Anti-Tetanus pre-booster (N = 93, 105) | 0.364 [0.308 to 0.431] | 0.504 [0.438 to 0.581]
  Anti-Tetanus post-booster (N = 93, 105) | 11.6 [9.71 to 13.9] | 24.7 [21.9 to 27.7]
  Anti-Pertusiss pre-booster (N = 89, 101) | 7.34 [6.22 to 8.64] | 6.82 [5.30 to 8.76]
  Anti-Pertusiss post-booster (N = 93, 105) | 128 [107 to 153] | 185 [149 to 229]
  Anti-FHA Pre-booster (N = 91,103) | 14.0 [11.3 to 17.3] | 2.21 [1.83 to 2.67]
  Anti-FHA Post-booster (N = 91,103) | 204 [179 to 233] | 158 [135 to 185]

3. Secondary Outcome: Number of Participants Reporting Solicited Injection Site Reaction or Systemic Reactions Following Vaccination With a Booster Dose of the DTaP-Hep B-PRP~T Combined Vaccine Concomitantly With Oral Polio Vaccine (OPV)
Description: Solicited injection site reactions: Pain, Erythema, and Swelling; Solicited systemic reactions; Pyrexia (temperature), Vomiting, Abnormal Crying, Drowsiness, Loss of Appetite, and irritability.
  Grade 3 reactions are defined as: Pain - cries when injected limb is moved; Erythema and Swelling - ≥ 5cm; Fever - rectal temperature ≥ 39.5ºC; Vomiting - ≥6 episodes per 24 hours; Crying - inconsolable crying for >3 hours; Somnolence - sleeping most of the time or difficulty to wake up; Anorexia - refuses ≥3 feeds; and Irritability - inconsolable.
Time Frame: Day 0 up to Day 7 after vaccination
Population: Safety was assessed on the safety analysis (intent-to-treat) population.
Measure: Number; unit: Participants
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Number analyzed (Participants) | 1230 | 613
Participants
  Injection site Pain post-vaccination | 411 | 216
  Grade 3 Injection site Pain post-vaccination | 10 | 1
  Injection site Erythema post-vaccination | 272 | 136
  Grade 3 Injection site Erythema post-vaccination | 7 | 3
  Injection site Swelling post-vaccination | 211 | 120
  Grade 3 Injection site Swelling post-vaccination | 7 | 4
  Extensive swelling of vaccinated limb | 0 | 0
  Pyrexia post-vaccination | 137 | 70
  Grade 3 Pyrexia post-vaccination | 0 | 3
  Vomiting post-vaccination | 53 | 33
  Grade 3 Vomiting post-vaccination | 3 | 0
  Crying post-vaccination | 98 | 58
  Grade 3 Crying post-vaccination | 0 | 0
  Somnolence post-vaccination | 114 | 73
  Grade 3 Somnolence post-vaccination | 0 | 0
  Anorexia post-vaccination | 97 | 53
  Grade 3 Anorexia post-vaccination | 2 | 3
  Irritability post-vaccination | 224 | 114
  Grade 3 Irritability post-vaccination | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 30 post-vaccination.
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Serious Adverse Events (participants affected / at risk) | 3/1230 | 0/613
Other Adverse Events (participants affected / at risk) | 411/1230 | 216/613
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: DTaP-Hep B-PRP~T + OPV (N=1230) | Group 2: Tritanrix-Hep B/ Hib™ + OPV (N=613)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Meningitis tuberculous (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: DTaP-Hep B-PRP~T + OPV (N=1230) | Group 2: Tritanrix-Hep B/ Hib™ + OPV (N=613)
Solicited injection site Pain (General disorders) | 411 | 216
Solicited injection site Erythema (General disorders) | 272 | 136
Solicited injection site Swelling (General disorders) | 211 | 120
Pyrexia (General disorders) | 137 | 70
Vomiting (Gastrointestinal disorders) | 53 | 33
Crying (Psychiatric disorders) | 98 | 58
Anorexia (Metabolism and nutrition disorders) | 97 | 53
Somnolence (Nervous system disorders) | 114 | 73
Upper respiratory tract infection (Infections and infestations) | 69 | 38
Irritability (Psychiatric disorders) | 224 | 114

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications